CLINICAL TRIAL: NCT03989778
Title: Efficacy of Vitamin D Supplementation and Metformin Compared to Metformin Alone for Improvement in Follicle Size of Infertile Females With Polycystic Ovary Syndrome: a Randomized Open Label Trial
Brief Title: Vitamin D and Polycystic Ovarian Syndrome (PCOS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Rehana Rehman, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 124
Record Dates: First submitted 2019-06-13; First posted 2019-06-18 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Infertility, Female; Infertility; Vitamin D Deficiency
MeSH Terms: conditions — Infertility, Female; Infertility; Vitamin D Deficiency | interventions — Vitamin D; Metformin

STUDY DESIGN:
Intervention Model Description: Infertile females with Polycystic Ovarian Syndrome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D supplement (Experimental): The intervention group will receive VD Cholecalciferol (D2) 50,000 I.U once weekly for 12 weeks, followed by 50,000 I.U once every fortnight for 24 weeks with the Metformin treatment as prescribed by the physician whereas
  Interventions: Drug: Vitamin D
- Control (No Intervention): control group will receive Metformin treatment during the study period.

INTERVENTIONS:
Drug: Vitamin D — Vitamin D supplementation
  Other Names: Metformin
  Arms: Vitamin D supplement

SUMMARY:
Primary Objectives:

To evaluate the efficacy of metformin and Vitamin D supplementation on serum insulin and serum androgen levels (Total testosterone, Steroid Hormone Binding Globulin, Free Androgen Index) levels compared metformin alone in infertile Poly cystic ovarian females of reproductive age group.

Secondary Objectives:

To measure change in endometrial thickness/number of follicles and follicular size by day 12 trans-vaginal ultrasound in the intervention group i.e. combination of metformin and vitamin D supplementation

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) as defined by "the presence of any two out of three criteria i.e. Oligo and/or anovulation, excess androgen activity and/or polycystic ovarian morphology on ultrasound", is a prevalent cause of female infertility. In the endocrine milieu of PCOS higher levels of insulin due to insulin resistance (IR) exert direct effects on the ovaries, release insulin-like growth factor 1 (IGF-1) from the liver and both then increase levels of testosterone. The resultant prevents the growth of ovarian follicles to acquire the required dimension for ovulation (i.e. > 10 mm) hence leading to anovulation and therefore subfertility. Vitamin D (VD) has found to be predominantly deficient in PCOS females, documented to cause IR giving rise to anovulatory cycles, hyperandrogenism and other significant features of PCOS. Therefore, we have hypothesized that treatment with VD in PCOS females can reduce IR, improve ovulation and signs of hyperandrogenism. Since Metformin is frequently prescribed for reducing IR and hence the treatment for anovulatory infertility in these females, we have planned to conduct an open label randomized control trial in PCOS infertile females who have vitamin D levels < than 25 ng/ml and are receiving Metformin therapy after ethical approval from Aga Khan University. The intervention group will receive VD Cholecalciferol (D2) 50,000 I.U once weekly for 12 weeks, followed by 50,000 I.U once every fortnight for 24 weeks with the Metformin treatment as prescribed by the physician whereas control group will receive Metformin treatment during the study period. We will compare change in number of dominant follicles (more than 10 mm) / endometrial thickness in both groups by Day 12 trans-vaginal ultrasound at the time of enrollment with scans done after 12 and 24 weeks. The other biochemical parameters [Total Testosterone, Steroid Hormone Binding Globulin, Free Androgen Index, Lipid Accumulation Product, Serum Insulin, Serum Triglycerides, Serum Calcium and Albumin] will be done at the time of recruitment in both the intervention and control groups and compared.

ELIGIBILITY:
Inclusion Criteria:

* Females with age range 18- 36 years, from all ethnic background having primary infertility with diagnosis of PCOS when at least 2 of these 3 elements are present: hyperandrogenism, chronic anovulation and polycystic ovaries and Vitamin D deficiency serum levels < 25 nmol/L

Exclusion Criteria:

exclusion criteria at baseline will be excluded from the study

* Females with secondary Infertility
* Hypercalcemia (plasma calcium concentrations> 2.65 mmol/L)
* Exclude women with Tuberculosis or other granulomatous disorders.
* Women receiving vitamin D replacement, oral contraceptives, hormonal replacement therapy, glucocorticoids, calcium supplementation, insulin-sensitizing drugs(incretin mimetic drugs, thiazolidinedione, sulfonylurea), lipid-lowering drugs or other drugs affecting insulin sensitivity or serum androgens (e.g., niacin, corticosteroids, beta-blockers, calcium channel blockers, thiazide diuretics), anti-epileptics, anti-retroviral, cholestyramine, anti-fungal, statins, H2 blockers, immunosuppressants, chemotherapeutic agents, antimicrobials (Rifampicin, isoniazid, hydroqychloroquin) or any other drug modifying lipid metabolism in the previous 3 months prior to study
* Women with congenital adrenal hyperplasia, Cushing's syndrome, androgen-secreting tumors, type 2 diabetes mellitus, renal, hepatic or thyroid disorders, hyperparathyroidism, malabsorption syndromes, Chronic Kidney Disease Hepatic failure, cystic fibrosis, vaginal bleeding of unknown etiology Women Those who had Bariatric surgery will also be excluded.

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-13 (Estimated)

PRIMARY OUTCOMES:
• Insulin levels | 24 weeks
  Decrease in insulin levels 60%
• serum androgen levels | 24 weeks
  Decrease in Serum Androgen levels

SECONDARY OUTCOMES:
Endometrial thickness | 24 weeks
  increase in endometrial thickness to 2mm
Lipid Accumulation Product | 24 weeks
  reduction in lipid accumulation product

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Rehana Rehman, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No